CLINICAL TRIAL: NCT04119752
Title: Effect of Curcumin on Microvascular Response and Tissue Oxygenation in Older People
Brief Title: Effect of Curcumin on Microvascular Response and Tissue Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, Director, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 97055018.1.0000.5699
Record Dates: First submitted 2019-04-24; First posted 2019-10-08 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Risk Factor
Keywords: Curcumin; Microvascular responsiveness; Aging; Tissue oxygen saturation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Curcumin powder (Active Comparator): Curcumin powder - 10g
  Interventions: Dietary Supplement: Curcumin powder
- Placebo ( curcumin depleted) (Placebo Comparator): Placebo- sucralose -1g
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curcumin powder — 10g of curcumin powder
  Arms: Curcumin powder
Dietary Supplement: Placebo — 1g of sucralose
  Arms: Placebo ( curcumin depleted)

SUMMARY:
Aging has been associated with reduced bioavailability of nitric oxide(NO) and endotelial dysfunction.Curcumin, a phenolic compound present in the rhizomes of turmeric, possesses cardiovascular protective, anti-inflammatory and antioxidante properties.

The present study is evaluating the effects of ingestion of 10 g of curcumin supplementation (CUR) on microvascular responsiveness and tissue oxygen saturation in the elderly with cardiometabolic risks.Twenty eight older individuals have been submitted to 10 g of curcumin suplementation (CUR) or placebo (PLA) (sucralose). Microvascular responsiveness and tissue oxygen saturation have been measured 120 minutes after interventions.

DETAILED DESCRIPTION:
Aging has been associated with reduced bioavailability of nitric oxide(NO) and endotelial dysfunction.

Curcumin, a phenolic compound present in the rhizomes of turmeric, possesses cardiovascular protective, anti-inflammatory and antioxidante properties.

The present study is evaluating the effects of ingestion of 10 g of curcumin suplementation(CUR) on endothelial function and muscle oxygen saturation in the elderly at cardiometabolic risks.

The study is randomized, crossed-over, double blind and controlled by placebo.Twenty-eight volunteers have been recruted for the research. They will perform three visits in vascular dymamic laboratory, that is located at the Federal Universite of Rio de Janeiro , campus Macaé. Basic measures have been performed on the first visit: systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR), maximal voluntary contraction (MVC), endothelial function analysis, vascular responsiveness during rest ( TOV) and rhythmic handgrip exercise. On second and third visits, after 10 minutes period of quiet in rest , volunteers are submitted (SBP), (DBP) and (HR), MVC, blood and urine samples are drawn at baseline in order to analyse curcumin absorption and verify oxidative stress markers( vitamin C and malondialdehyde). Moreover , volunteers are submitted to 10 g of curcumin supplementation (CUR) diluted in 400 ml cold water or placebo (sucralose) that is offered in capsules ingested with 400 ml of water. Microvascular responsiveness and muscle oxygen saturation have been is measured 120 minutes after intervention.Urine and blood samples have been drawn again 20 minutes after exercise.

Before each visit, participants are instructed to fast 8 hours avoiding ingestion of high nitrate such as ( sausages, cheeses, dark green leaves, beets), polifenols foods ( tea, coffee, grape juice and cocoa) and curcumin based dressings(turmeric, curry, colorau). Also, participants have been instructed not practice plysical activities and not change food habits during the research period.

ELIGIBILITY:
Inclusion Criteria:

* Seniors,
* With two or more risk factors for cardiovascular disease:Dyslipidemia, visceral obesity, hypertension, diabetes mellitus 2 and others.

Exclusion Criteria:

* Smoking,
* Use of antioxidant drugs during the experiment period,
* Allergy to components of curcumin,
* With previous history of cancer, HIV,
* Neurodegenerative and osteomioarticular diseases.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Changes in microvascular reactivity | Changes from baseline at 120 minutes after nutritional intervention
  Microvascular reactivity will be evaluated by using a near-infrared spectroscopy device during a vascular occlusion test.
Changes in tissue oxygen saturation | Changes from baseline at 120 minutes after nutritional intervention
  Muscle and cerebral oxygen saturation will be evaluated by using a near-infrared spectroscopy device during exercise

SECONDARY OUTCOMES:
Changes in nitric oxide metabolites (plasma nitrate and nitrite) | Changes from baseline at 120 minutes after nutritional intervention
  Nitric oxide metabolites will be evaluated by plasma nitrate and nitrite by using a high-performance liquid chromatography system.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rezende, Principal Investigator — UFRJ -Campus Macaé
Locations (1):
- Central Coexistence of the Elderly, Macaé, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Rezende C, Oliveira GV, Volino-Souza M, Castro P, Murias JM, Alvares TS. Turmeric root extract supplementation improves pre-frontal cortex oxygenation and blood volume in older males and females: a randomised cross-over, placebo-controlled study. Int J Food Sci Nutr. 2022 Mar;73(2):274-283. doi: 10.1080/09637486.2021.1972411. Epub 2021 Sep 22. PMID 34551650